CLINICAL TRIAL: NCT04255979
Title: A Randomized, Double-blind, Placebo-controlled Single Dosing, Dose Escalation Phase I Clinical Trial to Investigate the Safety/Tolerability and Pharmacokinetics of HY209 After Intravenous Administration in Healthy Male Volunteers
Brief Title: A Study of HY209 in Healthy Male Volunteers for Sepsis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shaperon (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HY209-IV
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled single dosing, dose escalation
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): Single dose of HY209 0.1 mg/kg or placebo.
  Interventions: Drug: HY209
- Cohort 2 (Experimental): Single dose of HY209 0.2 mg/kg or placebo.
  Interventions: Drug: HY209
- Cohort 3 (Experimental): Single dose of HY209 0.4 mg/kg or placebo.
  Interventions: Drug: HY209
- Cohort 4 (Experimental): Single dose of HY209 0.8 mg/kg or placebo.
  Interventions: Drug: HY209
- Cohort 5 (Experimental): Single dose of HY209 1.6 mg/kg or placebo.
  Interventions: Drug: HY209
- Cohort 6 (Experimental): Single dose of HY209 3.2 mg/kg or placebo.
  Interventions: Drug: HY209

INTERVENTIONS:
Drug: HY209 — 6 Subjects will be assigned to drug (HY209) and 2 subjects will be assigned to placebo.
  Other Names: HY209-IV

SUMMARY:
A randomized, double-blind, placebo-controlled single dosing, dose escalation phase I clinical trial to investigate the safety/tolerability and pharmacokinetics of HY209 after intravenous administration in healthy male volunteers

DETAILED DESCRIPTION:
HY209, which is being developed for the treatment of sepsis, inhibits inflammation by promoting the differentiation and division of Myeloid-derived suppressor cells (MDSCs).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male aged from 19 to 45 at screening test
* BMI 18 kg/m2 ~ 27 kg/m2 at screening test
* Subjects found to be clinically healthy by medical history, physical examination, vital signs, electrocardiogram (ECG), and appropriate laboratory tests
* Those who must be capable of giving informed consent and willing to comply with all clinic visits and study-related procedures for the duration of study until study completion

Exclusion Criteria:

* Those who have a history of hypersensitivity or clinically significant hypersensitivity reactions to drugs (containing Taurodeoxycholate component, aspirin, antibiotics, etc.)
* Those who showed clinical symptoms suspected of acute infectious disease within 2 weeks before the first does, or whose body temperature (ear canal) measured at screening showed 38 ℃ or higher
* Those who have a clinically significant disease of liver, kidney, digestive, respiratory, endocrine, neurologic, blood/tumor, cardiovascular system history of those diseases
* Those who have a history of gastrointestinal diseases or surgery that may affect the absorption of the investigational drug
* Those who have a history of substance abuse or have tested positive for drugs of concern for misuse by urine drug screening
* Patients with the following blood pressure measured at the seat after resting for more than 5 minutes at the screening visit [Systolic blood pressure (SBP): < 90 mmHg or > 150 mmHg, Diastolic blood pressure (DBP): < 50 mmHg or > 90 mmHg]
* Those who participated in other clinical trials or bioequivalence within 6 months prior to the first dosing and received the drug
* Those who have donated whole blood within 2 months before the first dose or ingredient donation within 1 month or received blood transfusion within 1 month
* Those who have taken metabolic enzyme-induced and inhibitory drugs within 1 month before screening
* Those who consumed grapefruit / caffeine-containing foods within 3 days of the first dose and who cannot refrain from eating grapefruit-containing foods from 3 days before admission to discharge date
* Those who have taken specialty or herbal medicines within 2 weeks of the first dose or who have taken over-the-counter (OTC) within 1 week
* Caffeine overdose, alcohol overdose or oversmoker
* Those who have unusual eating habits or who are unable to eat the meals provided in this clinical trial
* Other investigator judged to be unsuitable as clinical subject

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) | Up to Day 6
  Number of subjects with abnormal laboratory values and/or adverse events that are related to treatment

SECONDARY OUTCOMES:
Maximum concentration (Cmax) of HY209 | Up to Day 2
  Maximum concentration of HY209 in plasma
Ratio of area under curve infinity (AUCinf) of HY209 | Up to Day 2
  Area under the plasma HY209 concentration-time curve over the time interval from 0 extrapolated to infinity
Ratio of area under curve last (AUClast) of HY209 | Up to Day 2
  Area under the plasma HY209 concentration-time curve over the time interval from 0 to the last quantifiable plasma concentration
Time of maximum concentration (Tmax) of HY209 | Up to Day 2
  Time of maximum concentration of HY209 in plasma
Terminal halif-life (t1/2) of HY209 | Up to Day 2
  Terminal half-life of HY209 in plasma

CONTACTS AND LOCATIONS:
Overall Officials: In-jin Jang, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No